CLINICAL TRIAL: NCT05451082
Title: Registry-based Study in Patients With Hepatitis D Virus (HDV) Infection in China
Status: Not yet recruiting | Type: Observational
Sponsor: Lai Wei (Other)
Responsible Party: Sponsor-Investigator, Lai Wei, Professor, Beijing Tsinghua Chang Gung Hospital
Organization: Beijing Tsinghua Chang Gung Hospital (Other)
Other Study IDs: 22201-4-02
Record Dates: First submitted 2022-06-26; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Hepatitis D
Keywords: hepatitis D virus
MeSH Terms: conditions — Hepatitis D

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Group Assignment

SUMMARY:
This is a retrospective, prospective, noninterventive, multicenter registry study. Patients diagnosed with HDV infection (based on positive HDV RNA) were included in this study and were followed up for at least 5 years to evaluate their disease progression and clinical outcomes (including death, liver transplantation, hepatocellular carcinoma [hcc], liver decompensation, and cirrhosis) during the 5-year follow-up period. All patients were followed up at least once a year after they were included in the study.

It was in 2016 HDV infection first reported in China. Since January 1, 2016, all patients diagnosed with HDV infection can be enrolled in this study and evidence confirming the diagnosis (including but not limited to HDV RNA test reports and medical records, etc.) must be delivered. The main test results (including serum HDV RNA, ALT, and tests to determine the presence of liver cirrhosis, decompensation of liver function, and liver cancer such as B-ultrasound and FibroScan) of these patients each year from diagnosis to enrollment should be collected and filled in the case report form (CRF).

Follow-up data of patients with serum anti-HDV positive and HDV RNA negative can be recorded and followed up on this platform, with informed consent of the patients is required. Patients whose serum HBV RNA turn positive during the follow-up period will be included in the follow-up cohort of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 or above, both sex;
* Evidence of a positive test for HDV RNA can be provided on or before the enrollment date;
* Able to sign written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HDV-infected individuals with a positive HDV RNA test result
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of death of patients infected with HDV during 5-year follow-up | 5 years
  HDV means hepatitis D virus
The incidence of liver transplantation of patients infected with HDV during 5-year follow-up | 5 years
  HDV means hepaitis D virus
The incidence of hepatocellular carcinoma of patients infected with HDV during 5-year follow-up | 5 years
  HDV means hepaitis D virus
The incidence of liver decompensation of patients infected with HDV during 5-year follow-up | 5 years
  liver decompensation means ascites, variceal bleeding, or hepatic encephalopathy
The incidence of cirrhosis of patients infected with HDV during 5-year follow-up | 5 years
  Patients who developed cirrhosis in the absence of cirrhosis at baseline by liver biopsy or noninvasive testing

SECONDARY OUTCOMES:
Demographic characteristics of HDV-infected individuals using baseline data | 1 year
  Demographic characteristics: age, sex, height, weight, nationality, main residence, economic level.
Epidemiological characteristics of HDV-infected individuals using baseline data | 1 year
  Risk factors for infection/possible route of infection, HDV genotype
Serum HDV RNA levels of patients infected with HDV | 5 years
  HDV means hepaitis D virus
Serum HBV DNA levels of patients infected with HDV | 5 years
  HBV means hepaitis B virus, HDV means hepaitis D virus
HBsAg concentration levels of patients infected with HDV | 5 years
  HBsAg means Hepatitis B surface antigen，HDV means hepaitis D virus
Serum alanine aminotransferase concentration levels of patients infected with HDV | 5 years
  HDV means hepaitis D virus
Serum total bilirubin concentration levels of patients infected with HDV | 5 years
  HDV means hepaitis D virus
Serum albumin levels concentration levels of patients infected with HDV | 5 years
  HDV means hepaitis D virus
Child-Pugh scores of patients infected with HDV | 5 years
  The Child-Pugh classification is a universal scoring system of the degree of liver failure in patients with cirrhosis. Variables measured by this system include ascites, encephalopathy, serum albumin, bilirubin, and prothrombin time. Traditionally, the Child-Pugh class (A, B, or C) has been used as a predictive index for operative mortality rate in adult patients undergoing portosystemic shunting procedures. The estimated 1- and 5-year survival rates are 95% and 75% for patients with Child-Pugh class B, and 85% and 50% for patients with Child-Pugh class C.
The incidence of death of chronic HDV-infected patients with persistently normal ALT | 5 years
  HDV means hepaitis D virus, ALT means alanine aminotransferase
The incidence of liver transplantation of chronic HDV-infected patients with persistently normal ALT | 5 years
  HDV means hepaitis D virus, ALT means alanine aminotransferase
The incidence of hepatocellular carcinoma (HCC) of chronic HDV-infected patients with persistently normal ALT | 5 years
  HDV means hepaitis D virus, ALT means alanine aminotransferase
The incidence of liver decompensation of chronic HDV-infected patients with persistently normal ALT | 5 years
  HDV means hepaitis D virus, ALT means alanine aminotransferase
The incidence of cirrhosis of chronic HDV-infected patients with persistently normal ALT | 5 years
  HDV means hepaitis D virus, ALT means alanine aminotransferase
The proportion of patients with HDV RNA negative conversion of patients receiving antiviral therapies | 5 years
  HDV RNA negative conversion means HDV RNA< lower limit of quantification（LLOQ）
The proportion of patients with a >2lg IU/mL HDV RNA decline of patients receiving antiviral therapies | 5 years
  The proportion of patients with a HDV RNA decrease of greater than 2log IU/mL
Changes in serum HDV RNA during treatment and after discontinuation | 5 years
  HDV means hepatitis D virus
The proportion of patients with ALT normalization of patients receiving antiviral therapies | 5 years
  ALT means alanine aminotransferase，ALT normalization means ALT <ULN
Combined response rate of patients with antiviral therapy | 5 years
  Combined response means HDV RNA <LLOQ and ALT<ULN
Number of patients with abnormal laboratory values and/or adverse events that are related to antiviral treatment | 5 years
  Number of patients with adverse events, sever adverse events, abnormal laboratory parameters, and drug combinations

CONTACTS AND LOCATIONS:
Locations (1):
- Bejing Tsinghua Changgung Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR

REFERENCES:
- [Background] Lok AS, Negro F, Asselah T, Farci P, Rizzetto M. Endpoints and New Options for Treatment of Chronic Hepatitis D. Hepatology. 2021 Dec;74(6):3479-3485. doi: 10.1002/hep.32082. Epub 2021 Sep 16. No abstract available. PMID 34331781
- [Background] Rizzetto M, Hamid S, Negro F. The changing context of hepatitis D. J Hepatol. 2021 May;74(5):1200-1211. doi: 10.1016/j.jhep.2021.01.014. Epub 2021 Jan 20. PMID 33484770